CLINICAL TRIAL: NCT06999538
Title: Real-life Performance Evaluation of the LiFlow X-ray Platform
Acronym: LiFE
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49RC25_0203
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Solid Cancers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Radiologist interpretation — two interpretations (with and without Liflow, oncology imaging tool).

SUMMARY:
The thoraco-abdomino-pelvic (TAP) scanner is crucial for assessing and monitoring solid cancers. However, advancements in scanner technology have led to a significant increase in data volume, from 100 images per exam 20 years ago to 2,000 today. The rising number of cancer cases and treatments requiring closer monitoring further strain the workload, prolonging interpretation time and causing delays in therapeutic management and adjustments. The limited number of radiologists contributes to this saturation, increasing the risk of missing metastatic lesions, especially in the lungs, liver, bones, peritoneum, and lymph nodes. The RECIST 1.1 criteria, introduced 15 years ago for standardized follow-up, are useful but time-consuming to implement, resulting in only a small fraction of oncology CT reports using them.

DETAILED DESCRIPTION:
The LiFE study consists in retrospectively interpreting the TAP scans of patients who have agreed to take part in the study at two separate times, once without the LiFlow tool and once with it, at least 8 weeks after the scan date. To avoid any memory effect, a washout period of 8 weeks will be observed between these two interpretations. The study will involve 10 radiologists and 400 patients. Each scan will be interpreted twice by the same doctor (with and without the LF tool). During the second retrospective interpretation, the radiologist will assess the impact of of the additional lesions discovered by LiFlow on the patient's therapeutic management. The notion of change in management is defined by a change in treatment, such as a change in surgical technique, a change in chemotherapy or an indication for a treatment not initially planned. In addition, for these lesions, a gold standard will be obtained (an opinion from one or two other radiologists and/or other characterization imaging and/or biopsy/histology and/or follow-up of the lesion).

The aim of the study is to validate the time saved on interpretations and reports, and to improve the accuracy of TAP scan interpretation.

ELIGIBILITY:
Inclusion Criteria:

* TAP (thoraco-abdomino-pelvic) scans
* Age > 18 years

Exclusion Criteria:

* Examination of imperfect quality due to movement or breathing,
* Inability to inject contrast medium or incomplete injection
* refusal to use data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients treated for solid cancer
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Time elapsed between opening and closing, oncology interpretation completed, of the same file interpreted | 1 day

SECONDARY OUTCOMES:
Number of additional relevant lesions discovered | Day 1
Duration recorded for examinations with no relevant lesions and pathological examinations | Day 1
Recorded times for initial and follow-up examinations | Day 1
Location and size of lesion(s) on report and nature of primary tumor in patient file | Day 1
Number of lesions detected | Day 1
  relevant or doubtful lesions by reading with or without Liflow
Number of lesions whose discovery would have led to a change in treatment | day 1
  change in surgical technique, change in chemotherapy, indication of a treatment not initially planned
Number of lesions not retained | day 1

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Aube, Study Chair — University Hospital, Angers

IPD SHARING:
Plan to Share IPD: Undecided